CLINICAL TRIAL: NCT03465293
Title: Does Mechanical Bowel Preparation Destabilise the Gut Microbiota and Provide a Window of Opportunity in Which to Influence the Re-establishing Microbiota in Diverticulosis?
Brief Title: Influence of Mechanical Bowel Preparation on GI Microbiota
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Reading (Other)
Collaborators: Royal Berkshire Hospital (Unknown)
Responsible Party: Principal Investigator, Marie Lewis, Dr, University of Reading
Other Study IDs: FNSML1
Record Dates: First submitted 2018-03-07; First posted 2018-03-14 (Actual); Last update posted 2018-03-14 (Actual); Status verified 2018-03

CONDITIONS: Diverticulosis, Colonic; Microbiota
Keywords: Symptomatic diverticulosis; Microbiota; Bowel preparation
MeSH Terms: conditions — Diverticulosis, Colonic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Stool and urine will be taken for analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- SUDD post-menopausal female: Post-menopausal women with non-specific left side pain and altered bowel habit who are having mechanical bowel preparation for a colonoscopy
  Interventions: Other: Bacterial composition and activity after bowel preparation

INTERVENTIONS:
Other: Bacterial composition and activity after bowel preparation — Bacterial composition and activity and patient's symptoms will be assessed pre and post bowel preparation taken as part of the preparation to have a pre-planned colonoscopy

SUMMARY:
The mechanical bowel preparation (BP) used to clean the colon prior to colonoscopy frequently results in a significant but temporary reduction in patient's symptoms for a number of bowel disorders including symptomatic uncomplicated diverticular disease. The cause of this improvement is unknown.

We hypothesise that changes to the gut microbial population (microbiota) are responsible for this improvement and that the repopulation of the GI tract with bacteria following colonoscopy results in a return of their normal symptoms. This pilot study will test this in a preliminary way by examining the stool, urine and blood of patients before and after bowel preparation to detect any destabilising effect that BP has on the gut microbiota and to what extent the microbiota repopulates at 3 months If the hypothesis is proven, this study will show that BP generates a 'window of opportunity' in which to influence the subsequent re-establishment of the microbiota. This is with the eventual aim of correcting potential dysbiosis and preventing the progression of symptomatic uncomplicated diverticular disease (SUDD).

DETAILED DESCRIPTION:
The mechanical bowel preparation (BP) procedure, which directly precedes colonic endoscopy, results in a significant reduction in reported symptoms for several bowel disorders (eg irritable bowel syndrome (IBS )), but as yet, there is little research-based supporting evidence. This proposal will use a robust experimental design to explore both the composition of the microbiota, and importantly, its metabolic activity to assess interactions with human hosts following BP. The aim of this pilot study is to generate data demonstrating the destabilising effects of BP on both the composition and metabolic activity of the gut microbiota.

If the hypothesis is proven, this study will show that BP generates a 'window of opportunity' in which to influence the subsequent re-establishment of the microbiota. This is with the eventual aim of correcting dysbiosis and preventing the development of symptomatic uncomplicated diverticular disease in patients with diverticulosis.

Background Diverticular disease, characterised by weakness of the supporting connective tissue of the wall of the colon leading to the formation of diverticula1, is somewhat neglected and does not receive scientific attention that other inflammatory gut disorders have. Despite this condition affecting 50% of our aging population, approximately 1/5 of which will develop debilitating symptomatic uncomplicated diverticular disease (SUDD)2, there is a paucity of knowledge in this field.

The factors determining the transition from asymptomatic diverticulosis to SUDD are unclear. However, the gut microbiota has been implicated in a recent small-scale study which correlated diverticulosis with depletion of Clostridium cluster IV. Clostridium cluster IX, Fusobacterium and Lactobacillaceae, all of which can exert an anti-inflammatory effects. Patients who present with left-side non-specific abdominal pain and diarrhoea are assessed by colonic endoscopy. A small-scale study showed that this procedure also resulted in a significant reduction in Lactobacillaceae in the control population after 1 month (n=10).

BP is received 14 and 20 hours prior to colonoscopy and involves oral administration with a variety of stimulant laxatives (eg Moviprep - polyethylene glycol) resulting in severe diarrhoea and complete clearance of faecal matter from the bowel. It is likely that this BP is implicated in any reduction in reported symptoms as opposed to the endoscopic procedure itself, although putative underlying mechanisms have yet to be identified.

Hypothesis: Bowel preparation for endoscopy will destabilise the gut microbiota in patients with diverticulosis. Re-establishment of this microbiota follows an altered developmental trajectory resulting in sustained changes to the composition of the microbiota. Furthermore, these observed changes will have functional consequences as identified through altered metabolic interactions at the microbe-host interface.

Aims and objectives:

1. Quantify sustained observational changes which occur within the functional groups of the gut microbiota following BP (HTP FISHflow technology).
2. Functional consequences of such changes to host metabolism, host-microbe co-metabolism and short chain fatty acid production will be assessed (nuclear magnetic resonance spectroscopy and gas chromatography respectively).
3. Statistical data integration techniques will identify links between the altered microbiota and metabolic profiles to begin to determine the mechanisms underlying the influence of the gut microbiota in diverticulosis .
4. The outputs above will identify whether a 'window of opportunity' occurs following BP which could be exploited to rectify dysbiosis as a basis for a later larger-scale study.

Experimental design

In order to assess the effects of BP on the colonic microbiota in diverticulosis, post-menopausal women with mild non-specific left sided abdominal pain and diarrhoea, who have been referred to the colorectal unit at the Royal Berkshire Hospital , will be recruited by the applicants (KT, PC). Patients who have not received antibiotics in the previous 3 months will complete a questionnaire to assess gastrointestinal symptoms, which will be based on those used in our previous human Irritable Bowel Syndrome (IBS) trials. Urine will be collected at t=0 (before BP), t=2d (24h after BP), t=8d (1 week after BP) and t=3 months (when recalled to the hospital). Faeces will be collected at the same timepoints except t=2d, instead the first void following BP will be requested. Patients are sent oral BP by post or collect them from the endoscopy unit, and we will exploit this to deliver faecal sample pots. Samples will be provided either at the hospital and immediately frozen, or patients will be asked to freeze and bring with them to their appointment . Later samples (t-8d, t=3 months), will be kept frozen at home then collected by University of Reading staff once both samples have been collected. Upon collection, patients will be provided with the questionnaire (and self-addressed envelope) to allow comparison of their symptoms 2 weeks and 3 months post BP with those reported beforehand (t=0).

ELIGIBILITY:
Inclusion Criteria:

* Suspected symptomatic uncomplicated diverticular disease
* Requires colonoscopy for investigation of symptoms

Exclusion Criteria:

* Under 18yo
* Previous bowel resection
* Antibiotics use in the last 6 months
* Medical condition precluding colonoscopy

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Post-menopausal women with non-specific left side pain and an altered bowel habit who are due to be investigated by colonoscopy
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2018-05-01 (Estimated); Primary Completion 2018-10-01 (Estimated); Study Completion 2019-04-30 (Estimated)

PRIMARY OUTCOMES:
Composition of the colonic microbiota pre and post bowel preparation | 6 months
  Quantify sustained observational changes which occur within the functional groups of the gut microbiota following BP (HTP FISHflow technology)
Activity of the microbiota pre and post bowel preparation | 6 months
  Functional consequences of observed changes to host metabolism, host-microbe co-metabolism and short chain fatty acid production. This will be assessed by NMR spectroscopy and gas chromatography respectively

CONTACTS AND LOCATIONS:
Overall Officials: Marie Lewis, PhD, Principal Investigator — Reading University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Drago L, Toscano M, De Grandi R, Casini V, Pace F. Persisting changes of intestinal microbiota after bowel lavage and colonoscopy. Eur J Gastroenterol Hepatol. 2016 May;28(5):532-7. doi: 10.1097/MEG.0000000000000581. PMID 27015015
- [Result] Lozupone CA, Stombaugh JI, Gordon JI, Jansson JK, Knight R. Diversity, stability and resilience of the human gut microbiota. Nature. 2012 Sep 13;489(7415):220-30. doi: 10.1038/nature11550. PMID 22972295
- [Result] Merrifield CA, Lewis MC, Claus SP, Pearce JT, Cloarec O, Duncker S, Heinzmann SS, Dumas ME, Kochhar S, Rezzi S, Mercenier A, Nicholson JK, Bailey M, Holmes E. Weaning diet induces sustained metabolic phenotype shift in the pig and influences host response to Bifidobacterium lactis NCC2818. Gut. 2013 Jun;62(6):842-51. doi: 10.1136/gutjnl-2011-301656. Epub 2012 Jun 3. PMID 22661492